CLINICAL TRIAL: NCT01561768
Title: A Phase 2 Randomized, Observer-Blind, Dose-Ranging Study to Evaluate the Immunogenicity and Safety of Quadrivalent Seasonal Virus-Like Particle (VLP) Influenza Vaccine (Recombinant) in Healthy Young (18-64) Adults
Brief Title: A Study to Evaluate the Immune Response and Safety of a Seasonal Virus-Like Particle Influenza Vaccine in Healthy Young Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NVX 778.S205
Record Dates: First submitted 2012-03-02; First posted 2012-03-23 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Experimental)
  Interventions: Biological: Novavax Quadrivalent vaccine
- Group 2 (Experimental)
  Interventions: Biological: Novavax Quadrivalent vaccine
- Group 3 (Experimental)
  Interventions: Biological: Novavax Quadrivalent vaccine
- Group 4 (Experimental)
  Interventions: Biological: Novavax Trivalent vaccine
- Group 5 (Experimental)
  Interventions: Biological: cTIV

INTERVENTIONS:
Biological: Novavax Quadrivalent vaccine — Quadrivalent VLP vaccine: low dose; intramuscular injection, deltoid
  Arms: Group 1
Biological: Novavax Quadrivalent vaccine — Quadrivalent VLP vaccine: medium dose; intramuscular injection, deltoid
  Arms: Group 2
Biological: Novavax Quadrivalent vaccine — Quadrivalent VLP vaccine: high dose; intramuscular injection, deltoid
  Arms: Group 3
Biological: Novavax Trivalent vaccine — Trivalent Dose; intramuscular injection, deltoid
  Arms: Group 4
Biological: cTIV — Preconfigured dose; intramuscular injection, deltoid
  Arms: Group 5

SUMMARY:
The purpose of this study is to determine the immune response of three dose levels of the Novavax Quadrivalent vaccine in healthy young adults (18-64). The study is broken down into 5 treatment groups. Each group will enroll 100 subjects, for a total of 500 subjects. Group 1-3 will receive one of three dose levels of the Novavax Quadrivalent vaccine, Group 4 will receive a dose of the Novavax Trivalent vaccine, and Group 5 will receive a commercially available trivalent influenza vaccine (TIV). The study will also evaluate the safety and tolerability of the Novavax Quadrivalent vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or females, 18-64 years of age
2. Willing and able to give informed consent prior to study enrollment
3. Able to comply with study requirements
4. Women who are not post-menopausal (≥ 50 years of age and at least one year post last menses) or surgically sterile must have a negative urine pregnancy test at vaccination; will be advised through the Informed Consent process to avoid becoming pregnant over the duration of the study, and must assert that they will employ an effective form of birth control for the duration of the study. Acceptable forms of birth control are: credible history of abstinence from heterosexual activity, hormonal contraceptives (oral, injectable, implant, patch, ring), double-barrier contraceptives (condom or diaphragm, with spermicide), and intrauterine device (IUD)

Exclusion Criteria:

1. Participation in research involving investigational product (drug/biologic/device) within 45 days before planned date of first vaccination
2. History of a serious reaction to prior influenza vaccination, known allergy to constituents of licensed TIV (e.g., egg proteins) or polysorbate-80
3. History of Guillain-Barré Syndrome (GBS) within 6 weeks following a previous influenza vaccine
4. Received any vaccine in the 4 weeks preceding the study vaccination and any influenza vaccine within six months preceding the study vaccination
5. Any know or suspected immunosuppressive illness, congenital or acquired, based on medical history and/or physical examination
6. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
7. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study
8. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature >38.0°C on the planned day of vaccine administration)
9. Presence of chronic pulmonary (including asthma), cardiovascular (except hypertension), renal, hepatic, neurologic, hematologic or metabolic (including diabetes mellitus) disorders, which would include the potential subject in a "high-risk" category for influenza and/or its complications
10. Known disturbance of coagulation
11. Women who are breastfeeding or plan to become pregnant during the study
12. Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse
13. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of 3 dose levels of the Novavax Quadrivalent vaccine based on HAI responses | Day 21
Number of Solicited and Unsolicited Adverse Events for the Novavax Quadrivalent vaccine | 6 months

SECONDARY OUTCOMES:
Estimate capacity of the Novavax Quadrivalent vaccines to fulfill FDA criteria (immunogenicity) for all strains in healthy, young adults | Day 21
  Based on criteria of greater than or equal to 40% HAI seroconversion and greater than or equal to 70% of subjects with HAI titers greater than or equal to 1:40 post-vaccination.
Impact of including a fourth strain in the Novavax Quadrivalent vaccine on immune responses to other three strains | Day 21
  Based on comparison to a trivalent NovaFlu formulation tested at the 22.5ug of HA (per strain) dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Thomas, Ph.D., Study Director — Novavax
Locations (4):
- Australia (4):
  - CMAX, Adelaide
  - Emeritus Research, Melbourne
  - Linear Clinical Research, Perth
  - Holdsworth House, Sydney

REFERENCES:
- See also: Related Info — http://www.novavax.com